CLINICAL TRIAL: NCT03131011
Title: Body-image Satisfaction Following Permanent Black or Invisible UV Ink Tattoos for Localization of Adjuvant Radiotherapy Fields in Breast Cancer Patients
Brief Title: Body-image Satisfaction Following Permanent Black or Invisible UV Ink Tattoos
Acronym: SPOT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Reliable and consistent method of UV Tattoo application was not able to be achieved.
Sponsor: CancerCare Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RRIC 2017-011
Record Dates: First submitted 2017-04-13; First posted 2017-04-27 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer Female; Body Image Disturbance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - UV ink (Experimental): Radiotherapy tattoos will be applied using an invisible UV fluorescent ink that can only be detected while illuminated with a special ultraviolet flashlight.
  Interventions: Other: UV fluorescent ink
- Arm 2 - Black ink (No Intervention): Radiotherapy tattoos will be applied using standard black ink.

INTERVENTIONS:
Other: UV fluorescent ink — The use of UV tattoo ink results in a tattoo that is visible only under an ultraviolet light. Conventional black tattoo ink is replaced with UV ink for the application of radiotherapy "dot" tattoos. Handheld UV flashlights are used to make the tattoos visible for use during radiotherapy treatment set-up.
  Arms: Arm 1 - UV ink

SUMMARY:
A phase II prospective, randomized control trial assessing the impact of "invisible ink" ultra-violet (UV) tattoo ink versus conventional black tattoo ink for radiotherapy treatment localization on the quality of life of breast cancer patients undergoing adjuvant radiotherapy. The effect of tattoo type on quality of life will be measured objectively using the externally validated body-image satisfaction (BIS) scale as the primary outcome of interest, with secondary endpoints including: accuracy/reproducibility of radiotherapy setup using the invisible ink tattoos, resource impact requirements, and clinical feasibility. A sample size of 60 patients is planned (30 per study arm) with an anticipated accrual period of 18 months.

DETAILED DESCRIPTION:
Breast cancer patients ages 18-60 who are planned for adjuvant radiotherapy and who meet all inclusion/exclusion criteria will be offered voluntary participation in this trial. Recruitment will be open for approximately 18 months; it is anticipated that 1-2 patients will be recruited per week until the planned sample size is met. Participants will be stratified into three groups depending on their self-reported baseline Body-image satisfaction (BIS) score and will then be randomly allocated to receive conventional dark ink or UV fluorescent tattoos using permutated block randomization (4 patients per block) to ensure balance of BIS baseline average between study arms.

The investigators focus is to improve the current tattooing technique for breast cancer patients by introducing an alternate method that takes the patient's psychological perceptions of tattooing into account while first and foremost, continuing to guarantee that the current standard of accuracy in treatment delivery is maintained or improved. The investigators goal of decreasing the psychological effect of permanent radiotherapy tattoos aligns with CancerCare Manitoba's mission to improve the outcomes and quality of life for Manitobans with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female age 18-60.
* Histologically confirmed early stage invasive ductal or lobular carcinoma of a single breast (T1N0M0-T2N0M0) or DCIS/LCIS (TisNxMx or TisN0M0) of a single breast.
* Deemed fit to undergo adjuvant radiotherapy to their breast by their supervising radiation oncologist.
* Able to provide written informed consent.
* Must be willing to be contacted by e-mail and have a valid e-mail account to complete follow up self-reported body image scale questionnaires.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Intact skin at site of standard radiotherapy tattoos. Must have access to a computer and be able and willing to comply with requirements of the protocol.

Exclusion Criteria:

* History of any prior radiotherapy courses to the chest or abdomen.
* Metastatic disease.
* Node positive breast cancer.
* Bilateral breast cancer or bilateral DCIS/LCIS.
* Deep-inspiration breath hold radiotherapy technique.
* Unable or unwilling to comply with the requirements of the protocol as assessed by the study investigator or coordinator.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-04-23 (Actual)

PRIMARY OUTCOMES:
Change in Body-image scale score | Day 0, Week 3, Week 12
  Mean BIS scores at each time point will be calculated along with standard deviation and will be compared using the student t-test.

SECONDARY OUTCOMES:
Set-up Accuracy | Radiation Treatment week 1 (fractions 1, 2, 3) and Treatment week 2 (one fraction)
  Set-up accuracy will be assessed using orthogonal image sets from fractions 1, 2, 3 & one day treatment week 2 for each participant. Pre-imaging couch angle, vertical, longitudinal and lateral positions will be compared to the post-imaging values and evaluated based on our departmental couch adjustment tolerances for image-guided radiation therapy.
Resource Requirements (Tattooing procedure length) | Day 0 Simulation appointment, Radiation Treatment week 1 (fractions 1, 2, 3) and Treatment week 2 (one fraction)
  The average time(Min) it takes to complete the tattooing procedure during simulation will be collected and compared between the two arms.
Resource Requirements (Treatment set-up procedure length) | Day 0 Simulation appointment, Radiation Treatment week 1 (fractions 1, 2, 3) and Treatment week 2 (one fraction)
  The average time(Min) it takes to complete daily treatment set-up will be collected and compared between the two arms.
Radiation Therapist Evaluation Survey of UV Tattoo Method | Week 13
  Clinical practicability will be evaluated qualitatively through feedback from radiation therapists through a survey measuring their satisfaction with the UV tattooing method.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Kim, MD, MSc, Principal Investigator — CancerCare Manitoba; Erin V Toews, B.Sc., RTT, Principal Investigator — CancerCare Manitoba
Locations (1):
- CancerCare Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No